CLINICAL TRIAL: NCT05415189
Title: Lifetime Incidence and Socio-economic Implications of Mental Illness - a Nationwide Population-based Cohort Study
Brief Title: Lifetime Incidence and Socio-economic Implications of Mental Illness
Status: Completed | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: Lifetime incidence
Record Dates: First submitted 2022-06-07; First posted 2022-06-13 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Mental Illness
Keywords: Mental Illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with mental illness according to Danish health registers
  Interventions: Other: Not relevant
- Control individuals from the general population: Control individuals from the general population matched according to the data of diagnosis/ psychotropic medication, year of birth, sex and calendar year.
  Interventions: Other: Not relevant

INTERVENTIONS:
Other: Not relevant — This is a non-intervention cohort study

SUMMARY:
The purpose of the present study is to estimate the lifetime incidence of any mental disorder in a nationwide population-based register linkage study for the Danish population and to estimate the influence on socio-economic functioning.

DETAILED DESCRIPTION:
The purpose of the present study is to estimate the lifetime incidence of any mental disorder in a nationwide population-based register linkage study for the Danish population in total and according to gender and to estimate the influence on socio-economic functioning. The investigaters hypothesised that the lifetime incidence of any mental disorder is substantially higher than hitherto believed.

ELIGIBILITY:
Inclusion Criteria:

* The study was based on a randomly selected 1,500,000 sample of all persons who were registered in Statistics Denmark on the 1st of January 1995.

Exclusion Criteria:

* None

Ages: 1 Year to 110 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study was based on a randomly selected 1,500,000 sample of all persons who were registered in Statistics Denmark on the 1st of January 1995.
Sampling Method: Non-Probability Sample
Enrollment: 1500000 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Any psychiatric disorder or any psychotropic medication according to data in Danish nationwide registers | January 1, 1995 to December 31, 2020
  Cumulative incidens of any psychiatric disorder or psychotropic medication for any mental illness except sleep disorders, dementia and nicotine dependence in total and according to sex

SECONDARY OUTCOMES:
Diagnosis of any psychiatric disorder according to data in Danish nationwide registers | January 1, 1995 to December 31, 2020
  Cumulative incidence of a diagnosis of any psychiatric disorder in total and according to sex

OTHER OUTCOMES:
Socio-economic functioning in relation to individuals recorded with the primary outcome according to data in Danish nationwide registers | January 1, 1995 to December 31, 2020
  Socio-economic functioning

CONTACTS AND LOCATIONS:
Overall Officials: Lars V Kessing, Professor, Principal Investigator — Psychiatric Center Copenhagen
Locations (1):
- Psychiatric Center Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Data for this study is property of Statistic Denmark and the Danish Health Data Authority. The data are available from the authorities, but restrictions apply.

REFERENCES:
- [Derived] Kessing LV, Ziersen SC, Caspi A, Moffitt TE, Andersen PK. Lifetime Incidence of Treated Mental Health Disorders and Psychotropic Drug Prescriptions and Associated Socioeconomic Functioning. JAMA Psychiatry. 2023 Oct 1;80(10):1000-1008. doi: 10.1001/jamapsychiatry.2023.2206. PMID 37436730